CLINICAL TRIAL: NCT05227898
Title: Two-arm, Double-blind, Randomized Controlled Trial to Compare Efficacy of Two Digital Software Medical Devices as Interventions for Physical and Mental Health in Patients With Stage I-III Cancer
Brief Title: Virtual Trial to Compare Two Digital Therapeutics as Interventions for Physical and Mental Health in People With Cancer
Acronym: RESTORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Blue Note Therapeutics (Industry)
Collaborators: Curebase Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROT004
Record Dates: First submitted 2022-01-06; First posted 2022-02-08 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Cancer
Keywords: Breast Cancer; Colon/Rectal Cancer; Endometrial Cancer; Lymphoma; Leukemia; Lung Cancer; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Thyroid Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Lymphoma; Leukemia; Lung Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Attune™ (Active Comparator): Attune™ is a completely digital therapeutic intervention.
  Interventions: Device: Device: Attune™
- Cerena™ (Active Comparator): Cerena™ is a completely digital therapeutic intervention.
  Interventions: Device: Device: Cerena™

INTERVENTIONS:
Device: Device: Attune™ — People enrolled in the study use the app to complete ten informational sessions, each approximately 60-minute in length. The app also include guided exercises and other interactive opportunities.
  Arms: Attune™
Device: Device: Cerena™ — People enrolled in the study use the app to complete ten informational sessions, each approximately 60-minute in length. The app also include guided exercises and other interactive opportunities.
  Arms: Cerena™

SUMMARY:
This is a 2-arm randomized controlled study comparing how effective two therapeutic digital software devices are at improving anxiety and other indicators of psychological and physical health in patients with cancer. The study will be completely virtual, meaning participants can take part completely from home without visiting a clinic or study site.

The digital software devices, called called attune™ and cerena™, are designed to be used for approximately 12 weeks alongside oncology usual care regimens (medical, psychosocial). The study will enroll at least 352 stage I-III cancer patients with elevated anxiety symptoms who are currently receiving systemic treatment (radiation, chemotherapy, immunotherapy), have received systemic treatment within the last 6 months, or who have an established treatment plan that includes systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III cancer diagnosis
* Currently in active systemic treatment of chemotherapy, radiation or immunotherapy, have completed systemic treatment within the past 6 months, or have a treatment plan including planned systemic treatment.
* Are experiencing at least moderate anxiety
* 18 years of age or older
* Are fluent in English
* Have access to a smartphone (a mobile phone that performs many of the functions of a computer, typically having a touchscreen interface, internet access, and an operating system capable of running downloaded applications) or tablet that runs iOS or Android software, with cellular data service or wifi access.
* Willing to download software onto smartphone or tablet from Apple store or Android store

Exclusion Criteria:

* Systemic treatment plan includes only endocrine therapy.
* Treatment plan includes stem cell/bone marrow transplant.
* Currently participating in any other investigative CBT trial for treatment of anxiety or depression.
* Participant is unable to complete training, has cognitive deficits, more severe psychiatric conditions, lack of access to internet accessible device or psycho-social conditions (e.g., other social conditions, that would interfere with adherence to self-directed care), such that in investigator's opinion the participant would be unable to complete the study
* Recently completed use of Blue Note Therapeutics Covid Cancer Care Program or other Blue Note Therapeutics device or Blue Note Therapeutics-sponsored study
* Are experiencing severe levels of depression OR indicate suicidal risk (measured by surveys during screening for the study)
* Are experiencing anxiety below the required level (measured by a survey during screening for the study)
* Cancer diagnosis is melanoma, multiple myeloma, unstaged cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-02 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety | Baseline up to week 12
  The PROMIS-Anxiety (PROMIS-A) is a validated PRO consisting of 8 questions measuring anxiety symptoms. The change in PROMIS-A score over time will be assessed (reduction indicates reduced anxiety).

SECONDARY OUTCOMES:
Symptoms of depression | Baseline up to week 12
  The PROMIS-Depression (PROMIS-D) is a validated PRO consisting of 8 questions measuring depression symptoms. The change in PROMIS-D score over time will be assessed (decrease indicates reduced depression).
Symptoms of emotional distress | Baseline up to week 12
  Change in PROMIS Emotional Distress; a composite of PROMIS-Anxiety and PROMIS-Depression over time (decrease indicates reduced emotional distress).
Positive and negative affect | Baseline up to week 12
  The Positive and Negative Affect Schedule Short Form (PANAS-SF) measures positive and negative affect. Change in PANAS-SF scores over time will be assessed (increase in Positive Affect Scale indicates increase in positive emotions and expression; decrease in Negative Affect Scale indicates decrease in negative emotions and expression).
Cancer-related symptoms of anxiety (thought intrusions) | Baseline up to week 12
  The Impact of Events Scale-Revised (IES-R) is used to assess subjective distress caused by a stressful life event. The change in the IES-R Intrusion subscale mean score over time will be assessed (decrease in Intrusion score indicates reduced intrusive symptoms related to a specific stressor).
Wellbeing and quality of life | Baseline up to Week 12
  The Functional Assessment of Cancer Therapy - General (FACT-G) is designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. The change in FACT-G scores over time will be assessed (a reduction in the FACT-G total score, derived from the subscale scores, indicates an increased health-related quality of life).
Global Improvement-Likert Scale | Baseline up to Week 12
  The Global Improvement-Likert Scale uses a Likert scale to assess participant self-perception of the level of improvement of their overall well-being, symptoms of anxiety, and symptoms of depression since they began the study.
Symptom-related distress | Baseline up to week 12
  The Rotterdam Symptom Checklist (RSCL) is measures health-related quality of life of cancer patients. This study uses the same Likert scale and a subset of the symptoms ("eye strain" and "headache") that are part of the Rotterdam Symptom Checklist with the addition of the symptom "finger cramping" to monitor for all potential device adverse effects.
Perceived stress | Baseline up to Week 12
  The Perceived Stress Scale (PSS) measures how different situations affect feelings and perceived stress. The change in PSS scores over time will be assessed (higher PSS scores indicate higher perceived stress).
Level of stress management skill and coping skill efficacy (PAM) | Baseline up to Week 12
  The Patient Activation Measure (PAM) is used to assess the knowledge, skills, and confidence to manage one's health. The change in PAM scores over time will be assessed (higher PAM scores indicate higher patient activation).
Level of stress management skill and coping skill efficacy (MOCS Part A) | Baseline up to Week 12
  The Measure of Current Status (MOCS) Part A measures self-perceived status for using coping skills. The change in MOCS Part A scores over time will be assessed (increase indicates greater confidence in skill use ability).
Non-specific (social) intervention effects | Baseline up to Week 12
  The Measure of Current Status (MOCS) Part B assesses non-specific intervention effects - feelings of normalcy vs. alienation, sense of cohesiveness with other patients, perceptions of care from persons around them, and a sense of being better off than other cancer patients. The change in MOCS Part B scores over time will be assessed (increase indicates greater non-specific intervention effects).
Benefit Finding | Baseline up to Week 12
  The Benefit Finding Scale (BFS) assesses the perception that positive contributions were made to one's life by the experience of being diagnosed with and treated for cancer. The change in BFS scores over time will be assessed
Safety of each digital product | Baseline up to Week 12
  Self-reported device related adverse events; 3-item Distress Assessment and Response Tool (DART) self-reported to monitor suicidality.
Usability of each digital product | Week 12
  mHealth App Usability Questionnaire (MAUQ) mean scores will be measured at end of study (higher scores indicate higher ease of use / easier to use applications).
Acceptability of each digital product | Week 12
  Net promoter score (NPS), an index ranging from -100 to 100 that measures willingness to recommend the digital products, will be measured at end of study.

OTHER OUTCOMES:
Healthcare utilization | Baseline up to Week 12
  Incidence of ER visits, hospitalization, 30-day readmission rates, and average LOS for hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Dianne M Shumay, Principal Investigator — Blue Note Therapeutics
Locations (1):
- Www.Restoreclinicaltrial.Com, San Francisco, California, United States

REFERENCES:
- [Derived] Taub CJ, Zion SR, Ream M, Ramiller A, Heathcote LC, Eich G, Mendelsohn M, Birckbichler J, Ganz PA, Cella D, Penedo FJ, Antoni M, Shumay DM. Cognitive behavioral digital therapeutic effects on distress and quality of life in patients with cancer: National randomized controlled trial. J Consult Clin Psychol. 2024 Nov;92(11):727-741. doi: 10.1037/ccp0000911. PMID 39621368
- [Derived] Zion SR, Taub CJ, Heathcote LC, Ramiller A, Tinianov S, McKinley M, Eich G, Penedo FJ, Ganz PA, Antoni M, Shumay DM. Effects of a Cognitive Behavioral Digital Therapeutic on Anxiety and Depression Symptoms in Patients With Cancer: A Randomized Controlled Trial. JCO Oncol Pract. 2023 Dec;19(12):1179-1189. doi: 10.1200/OP.23.00210. Epub 2023 Oct 20. PMID 37862670